CLINICAL TRIAL: NCT04215458
Title: Microbiota in Skin and Mucosa of Patients With Inflammatory Skin Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Ditte Marie Saunte, Senior Consultant, PhD, Zealand University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: REG-102-2019
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Fungal Infection; Inflammatory Skin Disease; Yeast Infection Skin
Keywords: fungal colonization; inflammatory skin disease; yeast infection in skin
MeSH Terms: conditions — Mycoses; Dermatitis | interventions — Specimen Handling

STUDY DESIGN:
Intervention Model Description: case-control study
Masking Description: The staff that analyses the samples will not know whether they come from patients or volounteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sample collection (Other): Collection of samples investigating for yeast colonization in either patients with inflammatory skin disease or healthy controls.
  Interventions: Other: sample collection (swap or tape strip)

INTERVENTIONS:
Other: sample collection (swap or tape strip) — collection of swap or tape strip to determine yeast colonization in skin

SUMMARY:
The pathogeneses of many inflammatory diseases are not completely understood, yet, dysregulation of the human microbiota is increasingly being investigated as a possible contributing factor. The human microbiota includes bacteria, archaea, viruses and fungi. In general, little is known about the fungal colonization in inflammatory skin diseases.

This study aims to examine the prevalence of microbiome in skin and oral mucosa of a variety of patients and healthy volunteers visiting the Dermatological outpatient clinic.

The study is designed as a case-control study comparing the incidence of colonization or infection in skin and oral mucosa of patients with different skin diseases and healthy volunteers.

Patients with selected skin diseases, staff at Zealand University Hospital in Roskilde, relatives to staff and students with relation to the Dermatologic Department will be asked to fill out a short questionnaire and have swaps taken from oral mucosa, as well as skin scrapings and tape strips from lesional skin (only patients) and non-lesional skin (all).

DETAILED DESCRIPTION:
Background and aim The pathogeneses of many inflammatory diseases are not completely understood, yet, dysregulation of the human microbiota is increasingly being investigated as a possible contributing factor. The human microbiota includes bacteria, archaea, viruses and fungi. In general, little is known about the fungal colonization in inflammatory skin diseases although Candida species in oral mucosa, skin and feces seem to be increased in patients with psoriasis and atopic dermatitis. Inflammation is also an important part of the pathogenesis in other skin diseases such as hidradenitis suppurativa, acne, vasculitis and inflammatory ulcers. Possibly, increased fungal colonization may be present in many inflammatory skin diseases, yet, this has not previously been investigated. Studies of inflammatory diseases involving other body areas such as systemic lupus erythematosus, Sjögren's disease, multiple sclerosis, and spondyloarthritis have also demonstrated increased colonization with Candida species. However, it is unclear, whether colonization with Candida is a cause or a result of inflammatory disease. Treatment of inflammatory diseases with systemic immune-modulating drugs or recurrent antibiotic therapy may also affect yeast colonization. Emergence of biological therapies that directly or indirectly modulates the Interleukin (IL) 17-pathway emphasizes the need for further knowledge, since the IL-17 pathway is involved in the defense against yeast infections in healthy individuals. Until now, investigations of yeast colonization have primarily focused on Candida and Malassezia. Whether other species of yeasts may be of interest is still uncertain.

This study aims to examine the prevalence of microbiome and infection in skin and oral mucosa of a variety of patients and healthy volunteers visiting the Dermatological outpatient clinic.

Methods Study execution The project is carried out as a collaboration between Dermatological Department, Roskilde University Hospital and Statens Serum Institut (SSI) under the leadership of primary investigator, Senior Doctor in Dermatology, PhD, Ditte Marie Lindhardt Saunte. The project is supported by Medical Doctor in Dermatology, PhD Elisabeth Hjardem Taudorf, Dermatological study nurse Helle Anette Jensen, and the established research group at the Dermatological Department. The samples will be analyzed at SSI at the Dpt. of bacteria, parasites, and fungi under PhD Henrik Vedel Nielsen and Head of Microbial Bioinformatics, Department of Bacteria, Parasites and Fungi, PhD Marc Stegger.

Study design A case-control study comparing the incidence of yeast colonization or infection in skin and oral mucosa of patients with different skin diseases and healthy volunteers. Patients with selected skin diseases, staff at Zealand University Hospital in Roskilde, relatives to staff and students with relation to the Dermatologic Department will be asked to fill out a short questionnaire and have swaps taken from oral mucosa, as well as skin scrapings and tape strips from lesional skin (only patients) and non-lesional skin (all).

Swaps will be examined at Dept. of Microbial Bioinformatics, Department of Bacteria, Parasites and Fungi, Statens Serum Institut. The subgroup of patients initiating systemic therapy for their skin disease at the first examination will be asked to repeat the questionnaire, swaps, skin scrapings and tape strips after approximately three months.

Clinical photos of lesional skin or mucosa will be taken and stored at a secure IT site (Sharepoint and in SP clinical report) after written consent.

Statistics Prevalence and Odds Ratios (OR) will be determined. With a two-sided significance level of 95%, a power of 80 %, an expected ratio of healthy controls vs. patients with skin disease of 0.5 and an expected OR of 2.73 a minimum sample size of 127 patients per skin disease and 64 healthy controls are needed. We aim to include approximately of 130 patients per skin disease. In total, a maximum of 700 individuals will be included, of which 70 will be healthy controls. Inclusion of patients with rare skin diseases may necessitate fewer patients in some groups.

Risks, side effects and drawbacks All samples consist of non-invasive mucosal swaps, skin scrapings or superficial tape strips which holds no risk of known adverse effects. It may be associated with minimal discomfort during sample collection and participants may use an additional 15 minutes of their time in order to receive information regarding the project. Apart from that, this project causes no known risks, side effects or drawbacks.

Biologic material Swaps from mucosal membranes and skin. There is no biobank involved in this project.

Economy The Dermatologic Department, Roskilde University Hospital provides sample materials and Department of Bacteria, Parasites and Fungi, Statens Serum Institute, Copenhagen analyzes the samples. Both departments cover their own expenses. The project is completely independent and does not receive financial support from third parties. None of the involved research workers receive payment for participation or has conflicts of interest related to the project.

Remuneration for trial participants Participants will not receive any remuneration or compensation related to study participation.

Recruitment of trial participants and informed consent Patients, relatives and staff associated to the Dermatologic Department in Roskilde will be asked to participate. Patients and relatives will be recruited during a routine visit to the clinic, while staff will be offered participation during a regular staff meeting. A private consultation will take place, where each participant will receive individual oral and written information about the project in a quiet atmosphere. The participant can bring a bystander and will be offered time for consideration. If requested, an extra interview with repeated possibility to bring a bystander will be provided. If a person wants to participate in the project and meet criteria for inclusion, informed consent will be signed, a short questionnaire filled out and samples will be collected during their regular outpatient visit or by individual appointment.

Publication of results Positive as well as negative results will be published in relevant international Scientific Journals and presented at Scientific meetings and congresses.

Research ethics Many patients, staffs and relatives will be asked to participate in this case-control study, spend a short amount of extra time during an appointment at the clinic and may experience minimal discomfort during collection of samples. In contrast, information about microbiome in different skin diseases may provide a completely new insight and form the basis for further studies to detect the possible causality between microbiome and inflammatory skin diseases. Thus, the potential small disadvantages for project participants can by far be justified by the large amount of new knowledge obtained.

ELIGIBILITY:
Inclusion Criteria:

* Legally competent women and men
* Age 18 years or older

Exclusion Criteria

* Actual systemic or topical antifungal therapy
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of yeast colonization | at baseline
  detection of possible yeasts on the skin

SECONDARY OUTCOMES:
subtyping the possible yeasts found on the skin | at baseline
  subtyping by microscopy, culture or MALDI

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital Roskilde, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT04215458/Prot_SAP_000.pdf